CLINICAL TRIAL: NCT04558658
Title: Evaluation of Neutrophil to Lymphocyte Ratio in Inflammatory Bowel Disease in Assiut University Hospitals
Brief Title: Neutrophil to Lymphocyte Ratio in Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Mohammed, Evaluation of neutrophil-to-lymphocyte ratio in inflammatory bowel disease in assuit university hospitals, Assiut University
Other Study IDs: N/L ratio in IBD activity
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: neutrophil to lymphocyte ratio
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Complete Blood Count — neutrophil to lymphocyte ratio

SUMMARY:
Detection of Inflammatory Bowel Disease activity by Using new measure : Neutrophil to lymphocyte ratio

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) has been a global healthcare problem with a sustained increasing incidence. It includes two major forms, Crohn's disease (CD) and ulcerative colitis (UC), which are distinct chronic bowel-relapsing inflammatory disorders (Gharagozloo et al., 2015). Ulcerative colitis (UC) is limitd to Mucosa and cause continuous bowel inflammation (Celikbilek et al., 2013) While Crohn disease is more complex because of its transmural inflammation and it is characterized by skip lesions, which are diseased sections of bowel next to uninvolved areas(Nishijima David L; Wisner, David H; Holmes, James F, 2016). The prevalence of IBD is highest in the second to third decade of life with another peak in the 60-70- year-old group.(Silva et al., 2016) Non-invasive tests, such as C reactive protein (CRP), erythrocyte sedimentation rate (ESR) and white blood cells (WBC) are therefore being increasingly recognized as important markers for initial diagnosis and disease activity detection.(Gao et al., 2015) In recent years, the neutrophil-to-lymphocyte ratio (NLR), calculated as total neutrophil count divided by total lymphocyte count, NLR represents two different immune pathways and can be easily derived directly from a standard blood test..(Argeny et al., 2018)

ELIGIBILITY:
Inclusion Criteria:

* patients with inflammatory bowel disease, diagnosed by endoscopy, clinical , biochemical correlation and histopathological biopsy

Exclusion Criteria:

* patients have :
* Appendicitis
* sigmoid diverticular disease
* Infectious colitis
* patients known to have cancer colon

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed IBD by endoscopy, clinical , biochemical correlation and histopathological biopsy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil to lymphocyte ratio in IBD | baseline
  Determination of the prognostic value of N/L ratio in patients with IBD as a non invasive measure of disease acitivity

REFERENCES:
- [Background] Argeny S, Stift A, Bergmann M, Mittlbock M, Maschke S, Yang Y, Chitsabesan P, Riss S. Prognostic value of preoperative neutrophil-to-lymphocyte ratio in Crohn's disease. Wien Klin Wochenschr. 2018 Jun;130(11-12):398-403. doi: 10.1007/s00508-018-1322-3. Epub 2018 Feb 12. PMID 29435759
- [Background] Celikbilek M, Dogan S, Ozbakir O, Zararsiz G, Kucuk H, Gursoy S, Yurci A, Guven K, Yucesoy M. Neutrophil-lymphocyte ratio as a predictor of disease severity in ulcerative colitis. J Clin Lab Anal. 2013 Jan;27(1):72-6. doi: 10.1002/jcla.21564. Epub 2013 Jan 4. PMID 23292894
- [Background] Gao SQ, Huang LD, Dai RJ, Chen DD, Hu WJ, Shan YF. Neutrophil-lymphocyte ratio: a controversial marker in predicting Crohn's disease severity. Int J Clin Exp Pathol. 2015 Nov 1;8(11):14779-85. eCollection 2015. PMID 26823804